CLINICAL TRIAL: NCT06873438
Title: A Study on the Safety and Effectiveness of Lactobacillus Delbrueckii Subsp. Bulgaricus LB42 in Improving Intestinal and Immune Functions
Brief Title: The Effect of Probiotics on the Improvement of Intestinal and Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20250304
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Intestinal and Immune Function Improved

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Lactobacillus delbrueckii subsp. bulgaricus LB42 (30 billion CFU/day, 3g) was administered daily for 8 weeks. Store in a cool and dry place.
  Interventions: Dietary Supplement: Probiotic group
- Placebo group (Placebo Comparator): Every day to give 3g dextrin intervention for 8 weeks. Store in a cool and dry place.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Probiotic group — The experimental phase of this study will last 8 weeks and each subject will receive 3 follow-up visits (week 0, week 4, week 8).
  Arms: Probiotic group
Dietary Supplement: Placebo group — The experimental phase of this study will last 8 weeks and each subject will receive 3 follow-up visits (week 0, week 4, week 8).
  Arms: Placebo group

SUMMARY:
Evaluate the effectiveness and safety of Lactobacillus delbrueckii subsp. bulgaricus LB42 as a food supplement compared to a placebo in improving intestinal and immune functions in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years
2. Willing to undergo 3 follow-up visits during the intervention period
3. Willing to provide 2 blood, urine, and stool samples during the intervention period
4. Willing to self-administer one of the probiotics/placebo once daily during the intervention period
5. Good eyesight, able to read and write, and can wear glasses
6. Have good hearing and be able to hear and understand all instructions during the intervention

Exclusion Criteria:

1. Suffering from digestive disorders, mainly gastrointestinal disorders (celiac disease, ulcerative colitis, Crohn's disease)
2. Has a severe neurological condition (epilepsy, stroke, severe head trauma, meningitis within the past 10 years, brain surgery, brain tumor, prolonged coma - excluding general anesthesia)
3. Has received/is receiving treatment for the following psychiatric disorders: alcohol/drug/substance abuse dependence, schizophrenia, psychosis, bipolar disorder
4. Take medication for depression or low mood
5. Suffering from internal organ failure (heart, liver, or kidney failure, etc.)
6. Radiotherapy or chemotherapy in the past
7. Surgery/procedure under general anesthesia within the past three years, or planned to undergo a procedure/procedure under general anesthesia within the next 3 months during this trial
8. Have had hepatitis (hepatitis B, hepatitis C), HIV or syphilis in the past

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change in the concentration of LL-37 in feces before and after intervention. | Week 0 and Week 8
  Detected by Enzyme-Linked Immunosorbent Assay (ELISA).

SECONDARY OUTCOMES:
Change in the composition of fecal microbiota before and after intervention. | Week 0 and Week 8
  Analyzed by 16s RNA sequencing.
Change in the concentration of calprotectin in feces before and after intervention. | Week 0 and Week 8
  Detected by Enzyme-Linked Immunosorbent Assay (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- Xu fei, Zhengzhou, Henan, China